CLINICAL TRIAL: NCT06605521
Title: To Evaluate the Efficacy and Safety of Ipsilateral Supraclavicular Lymph Node Dissection for Breast Cancer Patients: A Prospective, Multicenter, Non-interventionist Real World Study
Brief Title: To Evaluate the Efficacy and Safety of Ipsilateral Supraclavicular Lymph Node Dissection for Breast Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2023-122
Record Dates: First submitted 2024-05-06; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-02

CONDITIONS: Locally Advanced Breast Cancer
Keywords: Supraclavicular lymph node dissection; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Control Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subclavian lymph node dissection+radiotherapy group: Subclavian lymph node dissection+radiotherapy
  Interventions: Procedure: Subclavian lymph node dissection+radiotherapy
- Simple clavicular region radiotherapy group: Simple clavicular region radiotherapy
  Interventions: Procedure: Simple clavicular region radiotherapy

INTERVENTIONS:
Procedure: Subclavian lymph node dissection+radiotherapy — The patient grouping is determined jointly by the researchers and participants, and patients in Group A are selected for supraclavicular lymph node dissection and radiotherapy.
  Other Names: experimental group
  Groups: Subclavian lymph node dissection+radiotherapy group
Procedure: Simple clavicular region radiotherapy — If the patient chooses Group B treatment plan, they will receive simple clavicle area radiotherapy.
  Other Names: control group
  Groups: Simple clavicular region radiotherapy group

SUMMARY:
For newly diagnosed ISLNM breast cancer, on the basis of effective treatment of the new auxiliary system, the optimal local treatment of the supraclavicular region remains controversial. Although guidelines such as NCCN recommend simple clavicular radiation therapy, there are studies suggesting that supraclavicular lymph node dissection can improve prognosis, and many hospitals in China are still accustomed to performing supraclavicular lymph node dissection. Therefore, ipsilateral supraclavicular lymph node dissection is the first time to diagnose ipsilateral supraclavicular lymph node metastasis of breast cancer. The effectiveness and safety of (stage IIIc) treatment still require prospective research to confirm.This project is a prospective, multicenter, non-interference real world study. In the real world study, the investigators evaluated the efficacy and safety of ipsilateral supraclavicular lymph node dissection in the treatment of initially diagnosed ipsilateral supraclavicular lymph node metastasis breast cancer patients.

DETAILED DESCRIPTION:
For newly diagnosed ISLNM breast cancer, on the basis of effective treatment of the new auxiliary system, the optimal local treatment of the supraclavicular region remains controversial. Although guidelines such as NCCN recommend simple clavicular radiation therapy, there are studies suggesting that supraclavicular lymph node dissection can improve prognosis, and many hospitals in China are still accustomed to performing supraclavicular lymph node dissection. Therefore, ipsilateral supraclavicular lymph node dissection is the first time to diagnose ipsilateral supraclavicular lymph node metastasis of breast cancer. The effectiveness and safety of (stage IIIc) treatment still require prospective research to confirm.This project is a prospective, multicenter, non-interference real world study. In the real world study, the investigators evaluated the efficacy and safety of ipsilateral supraclavicular lymph node dissection in the treatment of initially diagnosed ipsilateral supraclavicular lymph node metastasis breast cancer patients.

The main endpoint of the study was recurrence free survival on the ipsilateral clavicle. The secondary study endpoint is disease-free survival; Ipsilateral supraclavicular relapse-free survival; Rregional lymph node relapse-free survival; Overall survival; Security; The incidence of upper limb lymphedema; Patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged ≤ 80 years old.
2. ECOG score 0-1 points;
3. Breast cancer meets the following criteria: histologically diagnosed as invasive breast cancer, known ER, PR, HER2, KI67 status, pathologically diagnosed as ipsilateral supraclavicular lymph node metastasis (both cytology and histopathology);
4. Estimated patient survival time exceeding three months;
5. No obvious contraindications for surgery or radiotherapy;
6. The researcher judged that they were able to comply with the research protocol.
7. Those who participate in other clinical trials (including intervention or non intervention studies) at the same time and are judged by the researchers not to affect the research protocol can be enrolled normally.
8. Voluntarily participate in this study and sign an informed consent form.

Exclusion Criteria:

1. Stage IV (metastatic) breast cancer;
2. Bilateral breast cancer;
3. Received radiotherapy and surgical treatment (excluding local puncture) for ipsilateral supraclavicular metastatic lymph nodes before enrollment;
4. History of breast cancer or other malignant tumors, but excluding cured cervical carcinoma in situ, skin basal cell carcinoma or skin squamous cell carcinoma;
5. Individuals with severe primary diseases such as cardiovascular, cerebrovascular, liver, and kidney that are difficult to tolerate surgery or radiation therapy;
6. Having a history of immunodeficiency, including HIV testing positive, or having other acquired or congenital immunodeficiency diseases, or having a history of organ transplantation;
7. Suffering from severe comorbidities or other comorbidities that may interfere with the planned treatment, or any other circumstances in which the researcher deems the patient unsuitable to participate in this study.

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: cT1-4N3M0 breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2027-04-04 (Estimated); Study Completion 2027-04-04 (Estimated)

PRIMARY OUTCOMES:
Intraclavicular recurrence free survival in group A patients | 5th year after surgery
  The time from surgery to ipsilateral supraclavicular fossa recurrence or last follow-up.

SECONDARY OUTCOMES:
Disease-Free Survival | 5th year after surgery
  The time from surgery to the occurrence of recurrence, metastasis, or last follow-up.
Intraclavicular recurrence free survival in group B patients | 5th year after surgery
  The time from surgery to ipsilateral supraclavicular fossa recurrence or last follow-up
Regional lymph node recurrence free survival in group A/B patients | 5th year after surgery
  The time from surgery to the occurrence of regional lymph node recurrence, metastasis, or last follow-up
Overall survival of patients in Group A/B | 5th year after surgery
  The time from surgery to patient death or last follow-up
Number of adverse events | through study completion, an average of 2 year
  Complications related to surgery and radiotherapy
The incidence of upper limb lymphedema in group A/B patients at 2 years after surgery | 2th year after surgery
  Measure the circumference using the circumference method, with the styloid process of the ulna as the starting point, spaced 10cm apart and measured up to 40cm.
Patient's quality of life | 2th year after surgery
  Evaluate using the EORTC-QLQ-C30 V3 （European Organization of Research and treatment of Cancer-Questionnaire of Life Quality-C30 Version 3）scale.EORTC-QLQ-C30 V3 is the core scale of the quality of life measurement system developed by the European Organization for Research and Treatment of Cancer (EORTC) for cancer patients. The original scores of each item in the scale need to be converted into standardized scores ranging from 0 to 100 using linear formulas. The higher the scores of each functional dimension, the better the functional status; The higher the score of the symptom scale and individual items, the more obvious the symptoms and the poorer the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: xiuchun Chen, Study Chair — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China